CLINICAL TRIAL: NCT02988414
Title: Diagnosis of Bacteremia/Septicemia by the Karius Sequencing-Based Infectious Disease Diagnostic Assay
Brief Title: Diagnosis of Bacteremia/Septicemia and Culture Negative Endocarditis by the Karius Sequencing-Based Infectious Disease Diagnostic Assay
Status: Completed | Type: Observational
Sponsor: Karius, Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: 005-CL-01
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2017-04

CONDITIONS: Bacteremia; Septicemia
Keywords: Sepsis; Infection; Culture; Sequencing; Non-invasive; NGS
MeSH Terms: conditions — Bacteremia; Sepsis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Staphylococcus aureus Infection: Patients with blood culture confirmed S. aureus bloodstream infections.
- Gram Negative Infection: Patients with blood culture confirmed Gram Negative bloodstream infecrions
- Endocarditis: Patients admitted for evaluation of acute endocarditis classified using the Duke Criteria.

SUMMARY:
Prospective study at Duke University Hospital comparing the Karius Infectious Disease Diagnostic Sequencing Assay to blood culture results in admitted patients with bacteremia/septicemia.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. A positive blood culture
3. A suitable residual blood sample collected within 24 hours of the positive blood culture OR
4. A blood sample obtained for the study obtain within 48 hours of the positive blood culture

For Endocarditis Cohort:

1. All criteria above must be met and patient is admitted to the hospital and evaluated for acute endocarditis classified per the Duke Criteria

Exclusion Criteria:

1. Inability to understand instructions and comply with study-related procedures
2. Any condition that in the opinion of the treating physician will prevent the subject from completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are at least 18 years of age, have been admitted to Duke University Hospital, and have a positive blood culture.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value, and negative predictive value of the Karius test compared with blood culture in patients with bacteremia/septicemia | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vance G Fowler, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided